CLINICAL TRIAL: NCT03451968
Title: Twenty Four Hours Amino Acid Metabolism in Fed Surgical Critically Ill Patients: a Stable Isotope Tracer Study.
Brief Title: Amino Acid Metabolism in Fed Surgical Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Texas A&M University (Other)
Responsible Party: Principal Investigator, Pierre Singer, Professor, Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0281-17-RMC
Record Dates: First submitted 2017-12-27; First posted 2018-03-02 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Metabolism and Nutrition Disorder
Keywords: amino acid; stable isotope; critical care
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- critically ill (Experimental): amino acid tracer injection for metabolism analysis The dose needed to be injected from the tracer element in the beginning of the study is a bolus of 16ml Amino acid tracer (non-radioactive).
  it is a single bolus, no other elements or drug will be administered.
  Interventions: Other: amino acid tracer injection for metabolism analysis
- control (Active Comparator): amino acid tracer injection for metabolism analysis The dose needed to be injected from the tracer element in the beginning of the study is a bolus of 16ml Amino acid tracer (non-radioactive) it is a single bolus, no other elements or drug will be administered.
  Interventions: Other: amino acid tracer injection for metabolism analysis

INTERVENTIONS:
Other: amino acid tracer injection for metabolism analysis — the intervention includes injecting stable amino acid tracers in order to evaluate differences in processing of amino acid in critically ill patients compared to a normal population.
  after injection 5 ml of blood will be drawn at time 0, 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180 minutes from the start of the study, a total of 14 blood samples (70 cc).

SUMMARY:
Introduction Sarcopenia is defined as progressive generalized loss of skeletal muscle mass, strength and function. Sarcopenia due to lack of physical activity is a known phenomenon and is usually observed as a normal part of aging or in certain diseases and pathogenic processes. Major associated factors causing development of sarcopenia may be summarized as interactions of environmental and hormonal factors, underlying diseases, activation of inflammatory pathways, mitochondrial dysfunction, reduced satellite cell numbers, and loss of neuromuscular junctions.

Intensive care acquired weakness (ICU-AW) known formerly as critical illness polyneuropathy, is a diagnosis that becomes more common as survival rates from long ICU hospitalization are more prevalent. It is characterized by a primary axonal degeneration, without demyelination, that typically affects motor nerves more than sensory nerves.

ICU-AW affects the limbs (particularly the lower extremities) in a symmetric pattern. Weakness is most notable in proximal neuromuscular areas (e.g., the shoulders and hip girdle). In addition, involvement of the respiratory muscles can occur and can impede weaning from mechanical ventilation.

The pathophysiological mechanisms of ICU-acquired weakness are believed to be multifactorial. Some suspected factors include dysfunctional microcirculation and hyperglycemia. It has been shown that tight glucose control in ICU patients reduces the risk for ICU-AW (although it has been associated with other adverse events). Sodium channels channelopathy is also a researched cause for ICU-AW. Muscle loss in the ICU are usually related to bedridden condition and lack of mobility, increase in ubiquitination and inadequate protein administration associated with large negative nitrogen balance. In addition mechanical ventilation contributes greatly to this problem. This has been particularly relevant in post trauma/surgical long stayer patients.

In the past years great progress was made in the investigation of protein balance, breakdown and synthesis using stable isotope tracers in various medical conditions. In a research performed in PICU (1-5) and ICU (6, 7) regarding the measurement of plasma amino acid during critical illness, stable phenylalanine, tyrosine leucine, arginine and citrulline isotope were used intravenously without any safety issue problem. Another study was performed on adults suffering from COPD with matched healthy adults, using stable isotopes of phenylalanine, tyrosine leucine, isoleucine and valine (8). During the study the isotopes were given parenterally as well as enterally. The study showed significant change in splanchnic extraction of various amino acids and higher turnover of BCAA in COPD patients. Using the theory that supplemental milk can compensate for the elevated turnover of BCAA in COPD patients, using the isotope analysis demonstrated that this theory was proven wrong and the conclusion was that alterations are present in BCAA metabolism despite normal plasma levels in normal weight COPD. Further research is needed to find a way to compensate for it. These studies and other recent studies (9-19) show us the safety regarding the use of stable isotope tracers whether IV or PO, while giving us the opportunity to assess the metabolism of amino acid in all sorts of pathological states.

Hypothesis & Aim of the study We think that based on current literature, there are important differences between critically ill patients and healthy population in the amino acid profile and distribution in the body as well as synthesis and breakdown.

The aim of the study is to measure these differences in long ICU stayers (above 7 days) admitted in the ICU after surgical/trauma injury, and to try and help aiming future treatment and research in this field.

ELIGIBILITY:
Inclusion Criteria:

Study population:

* 15 ICU critically ill patient hospitalized due to surgical/trauma injury.
* above 18 years old no upper limit.
* hospitalized at the ICU more than 7 days

Control group:

* 15 Healthy volunteers, over 18 years old no upper limit.
* the volunteers won't be dependent or subordinated to the research investigators

Exclusion Criteria:

1. patients under 18 years old
2. patients under TPN treatment prior to their admission to ICU
3. patients with chronic bowel disease (e.g Crohn's, celiac, short bowel)
4. any relation (e.g family member or assistant) to the study investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
The amount of each amino acid will be measured in mmol/liter | during 3 hours from injection
  In the study stable isotopes of amino acids will be injected, and afterward the amount of each amino acid will be checked in order to assess degradation and metabolism. Composite measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No